CLINICAL TRIAL: NCT01490567
Title: Donepezil Adjunctive Treatment for Cognitive Impairment in Schizophrenia
Brief Title: A Double-blind, Placebo-controlled Trial of Donepezil Adjunctive Treatment for Cognitive Impairment in Schizophrenia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, xiaofeng Guo, Principal Investigator, Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NSFC30900485; 201002003 (Other Grant/Funding Number: the R&D Special Fund for Health Profession in China)
Record Dates: First submitted 2011-11-09; First posted 2011-12-13 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Impaired Cognition; Schizophrenia
Keywords: Impaired Cognition Schizophrenia
MeSH Terms: conditions — Cognition Disorders; Schizophrenia | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): Subjects will be given with a dose of 5mg/day placebo. All drugs will be administered orally.
  Interventions: Drug: placebo
- donepezil (Active Comparator): Subjects will be given with a dose of 5 mg/day donepezil. All drugs will be administered orally.
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Donepezil — 5 mg/day
  Other Names: Donepezil hydrochloride
  Arms: donepezil
Drug: placebo — placebo 5mg/d
  Arms: placebo

SUMMARY:
The objective of the study was to study the effects of donepezil on cognition in patients with schizophrenia. The investigators conducted a 12-week, double-blind, placebo-controlled trial of donepezil as adjunctive treatment to antipsychotic drugs on patients with schizophrenia.

DETAILED DESCRIPTION:
The investigators conducted a 12-week, double-blind, placebo-controlled trial of donepezil as adjunctive treatment to antipsychotic drugs on patients with schizophrenia.The trial will be complete in 2012.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia as determined by the Structured Clinical Interview for DSM-IV Axis I Disorders-Clinician Version;
* Between 18 and 40 years of age;
* Duration of the illness must be longer than 2 year;
* Patient's current antipsychotic medication regimen must be stable;
* Must be in a stable living arrangement;

Exclusion Criteria:

* Patient has mental retardation or severe organic brain syndromes;
* Treatment with Electroconvulsive Therapy (ECT) within 6 months prior to screening;
* Has suicidal attempts or ideation or violent behavior within the last 12 months;
* Patient has a history of alcohol/drug dependence;

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Mean Change From Baseline in the Composite Score From the Cognition Assessment Battery After 12 Weeks of Treatment | 12 weeks

SECONDARY OUTCOMES:
Mean Change From Baseline in Cognition Assessment scores After 12 Weeks of Treatment | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Guo, doctor, Principal Investigator — Second Xiangya Hospital of Central South University
Locations (1):
- the Second Xiangya Hospital of Central South University, Changsha, Hunan, China